CLINICAL TRIAL: NCT04626232
Title: Monocentric Prospective Randomized Controlled Study Comparing the Sleeve Gastrectomy Technique With a Nissen Fundoplication Added to the Conventional Sleeve Gastrectomy Technique (N-Sleeve) in Morbidly Obese Patients
Brief Title: Comparison of the Sleeve Gastrectomy Technique With a Nissen Fundoplication Added to the Conventional Sleeve Gastrectomy Technique in Morbidly Obese Patients
Acronym: N'SLEEVE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: no inclusions
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RECHMPL20_0013
Record Dates: First submitted 2020-10-08; First posted 2020-11-12 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Severe Obesity; GERD; Bariatric Surgery Candidate; Morbid Obesity
Keywords: Obesity; GERD; Surgery
MeSH Terms: conditions — Obesity, Morbid; Gastroesophageal Reflux; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- N SLEEVE (Experimental): Monocentric, randomized, single-blind controlled trial, with 2 parallel arms (experimental technique versus surgical reference technique).
  Interventions: Procedure: N-SLEEVE technique
- SLEEVE (Other): The conventional sleeve gastrectomy technique consists of reducing the gastric capacity by removing 2/3 of the stomach by a vertical transection.
  Interventions: Procedure: SLEEVE

INTERVENTIONS:
Procedure: N-SLEEVE technique — The N-SLEEVE technique (figure 2) consists of creating a gastric total fundoplication (Nissen technique) before to perform the removal of 2/3 of the stomach (SLEEVE technique).
  Arms: N SLEEVE
Procedure: SLEEVE — SLEEVE Technique : Removal of 2/3 of the stomach
  Arms: SLEEVE

SUMMARY:
The purpose of this study is to evaluate the impact of the procedure (sleeve gastrectomy technique with a Nissen fundoplication (N-Sleeve) vs conventional sleeve gastrectomy technique

DETAILED DESCRIPTION:
Bariatric surgery is recognized as the only effective therapeutic weapon for morbidly obese patients. Gastro-Oesophageal Reflux Disease is very common (30-45% of cases) with serious consequences on the oesophageal mucosa. It could be an exacerbation of preoperative GERD symptoms or a "de novo" postoperative GERD. Medical treatment is usually effective but reoperation may be required to treat refractory GERD.GERD can lead to serious consequences on the oesophageal mucosa (esophagitis, Barrett's oesophagus, cancer). The conventional surgical treatment of GERD is fundoplication, which can be partial or total. The gastric fundus is wrapped around the oesophagus to strengthen the tone of the oesophageal sphincter. We hypothesize that the creation of a total anti-reflux fundoplication before performing LSG (Nissen + Sleeve = N-sleeve) could significantly reduce the postoperative GERD complication as compared with the standard LSG.

To evaluate the impact of the procedure N-Sleeve vs conventional sleeve gastrectomy technique on the rate of patient with GERD at 1, 6 and 12 months postoperatively. To evaluate the impact of the procedure (sleeve gastrectomy technique with a Nissen fundoplication (N-Sleeve) vs conventional sleeve gastrectomy technique during all the follow-up on the gastric fistula on the staple line, on the postoperative morbidity and mortality , on the evolution of weight loss, the excess weight loss, the BMI and the excess BMI loss during the follow-up. Evaluate the impact of these procedures on the quality of life of patients at baseline and 1, 6 and 12 months postoperatively. Evaluate the safety during all the follow-up.

•Methods: Monocentric, randomized, single-blind controlled trial, with 2 parallel arms. 144 patients. The target population is all adult patients with severe or morbid obesity, who underwent multidisciplinary care and having the criteria of 2009 HAS recommendations for bariatric surgery.

Presence of gastro-oesophageal reflux will be assessed by a composite criteria: consumption of Proton Pump Inhibitor and gastroscopy at baseline and 12-month.

The N-SLEEVE technique consists of creating a gastric total fundoplication before to perform the removal of 2/3 of the stomach.

This study may really lead to a change in terms of choice of first intention bariatric procedures.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form
* Subjects must be able to attend all scheduled visits and to comply with all trial procedures
* Subjects must be covered by public health insurance
* Contraception efficacy
* Subjects eligible for sleeve gastrectomy after multidisciplinary evaluation according to HAS 2009 criteria: BMI ≥ 40 kg / m² with failure of the dietary treatment for at least 1 year, or a BMI ≥ 35kg / m² with at least one co-morbidity that could be improved after surgery (hypertension, obstructive sleep apnea hypopnea syndrome (OSAHS) and other severe respiratory disorders, severe metabolic disorders (especially type 2 diabetes), debilitating musculoskeletal diseases, non-alcoholic steato-hepatitis (NASH))

Exclusion Criteria:

* Subject unable to read or/and write
* Planned longer stay outside the region that prevents compliance with the visit plan
* Current pregnancy
* Previous bariatric surgery (ring, vertical banded gastroplasty, sleeve gastrectomy or Gastric Bypass).
* BMI > 50 kg / m² for women and > 45kg / m² for men (dissecting the hiatus region can be a technical challenge in these cases).
* Barrett oesophagus and esophagitis stage III and IV.
* Funditis
* Long-term NSAIDs and/or corticosteroid therapy
* No affiliation at the French social security scheme.
* Major protected by law.
* Deprivation of liberty by judicial or administrative decision.
* Participation to another clinical research program.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2022-09-12 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Presence of gastroesophageal reflux disease | 12 months
  Gastroscopy is a standard endoscopic examination that examines the lining of the oesophagus and stomach. It can detect Helicobacter pylori and highlight the presence of:
  * Gastro-Oesophageal Reflux Disease
  * Gastritis
  * Esophagitis
  * Barrett's oesophagus
  * Hiatal hernia
  * Gastric tumor
  * Bile reflux
  * Incompetent cardia
Consumption of Proton Pump Inhibitor | 12 months
  The consumption of PPI, revealing the presence of GERD symptoms, will be recorded at each visit thanks a diary card.

SECONDARY OUTCOMES:
type of fistula Month 1 | Month 1
  The diagnosis is confirmed by conducting a CT with contrast medium opacification. 4 stages are defined I, II, III and IV. TDM will be realized only in case of suspicion of fistulas (fever, pain in the left shoulder, vomiting).
  The type, the severity and the time between the date of occurrence of fistula and the date of the surgery will be recorded at each visit.
severity of fistula Month 1 | Month 1
  The severity of fistula is classified depending on the classification of Montpellier 2013 (Nedelcu)
type of fistula Month 6 | Month 6
  The diagnosis is confirmed by conducting a CT with contrast medium opacification. 4 stages are defined I, II, III and IV. TDM will be realized only in case of suspicion of fistulas (fever, pain in the left shoulder, vomiting).
  The type, the severity and the time between the date of occurrence of fistula and the date of the surgery will be recorded at each visit.
severity of fistula Month 6 | Month 6
  The severity of fistula is classified depending on the classification of Montpellier 2013 (Nedelcu)
type of fistula Month 12 | Month 12
  The diagnosis is confirmed by conducting a CT with contrast medium opacification. 4 stages are defined I, II, III and IV. TDM will be realized only in case of suspicion of fistulas (fever, pain in the left shoulder, vomiting).
  The type, the severity and the time between the date of occurrence of fistula and the date of the surgery will be recorded at each visit.
severity of fistula Month 12 | Month 12
  The severity of fistula is classified depending on the classification of Montpellier 2013 (Nedelcu)
Postoperative morbidity Month 1 | Month 1
  Assessed by the type of postoperative complication
Postoperative morbidity Month 6 | Month 6
  Assessed by the frequency of each type of postoperative complication
Postoperative morbidity Month 12 | Month 12
  Assessed by the severity of each type of postoperative complication
Weight loss Month 1 | Month 1
  The evolution of the weight of the patients will be assessed by measuring their weight in kilograms on the same scale at each visit in the digestive surgery service. The height (in meter) will be assessed at baseline in the digestive surgery service. The BMI will be calculated at each visit.
Weight loss Month 6 | Month 6
  The evolution of the weight of the patients will be assessed by measuring their weight in kilograms on the same scale at each visit in the digestive surgery service. The height (in meter) will be assessed at baseline in the digestive surgery service. The BMI will be calculated at each visit.
Weight loss Month 12 | Month 12
  The evolution of the weight of the patients will be assessed by measuring their weight in kilograms on the same scale at each visit in the digestive surgery service. The height (in meter) will be assessed at baseline in the digestive surgery service. The BMI will be calculated at each visit.
mortality Month 1 | Month 1
  number of death
mortality Month 6 | Month 6
  number of death
mortality Month 12 | Month 12
  number of death
Quality of Life Month 1 : SF 12 | Month 1
  Quality of life will be assessed by the self-questionnaire SF12
Quality of Life Month 6 : SF 12 | Month 6
  Quality of life will be assessed by the self-questionnaire SF12
Quality of Life Month 12 : SF 12 | Month 12
  Quality of life will be assessed by the self-questionnaire SF12
Serious adverse event Month 1 | Month 1
  number and type of adverse events
safety Month 6: number and type of adverse events | Month 6
  number and type of adverse events
safety Month 12: number and type of adverse events | Month 12
  number and type of adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Montpellier, Montpellier, France